CLINICAL TRIAL: NCT01974193
Title: Prevention of Pelvic Lymphocele by Floseal During Pelvic Lymphadenectomy for Gynecologic Cancer: a Pilot Study
Brief Title: Prevention of Pelvic Lymphocele by Floseal During Pelvic Lymphadenectomy for Gynecologic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Yun Hwan KIM, Assistant Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: BFL01
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Floseal (Experimental): application of floseal to one side of pelvis after pelvic lymphadenectomy
  Interventions: Drug: Floseal
- Control (No Intervention): counter-site of pelvis; no intervention after pelvic lymphadenectomy

INTERVENTIONS:
Drug: Floseal — application of floseal on intervention arm
  Arms: Floseal

SUMMARY:
Pelvic lymph node dissection (PLND) is an important step in the surgical staging and treatment of gynecologic malignancies.

Sometimes, complicated lymphoceles after PLND often delay adjuvant treatment including chemotherapy and radiation therapy, which potentially affects the success of cancer treatment.

A number of surgical techniques have developed, but failed to reduce the incidence of pelvic lymphoceles after PLND.

The investigators hypothesized that floseal can prevent lymphoceles in patients with gynecologic cancer who has undergone PLND.

The investigators designed prospective randomized controlled study as a pilot study.

The investigators will randomly apply floseal to one side of pelvis after bilateral PLND, and observe the occurence of pelvic lymphoceles after 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer patients who need laparotomic bilateral PLND

Exclusion Criteria:

* Incomplete PLND which can influence the occurrence of lymphocele (surgeon's decision)

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of pelvic lymphocele | 6 month
  Frequency of ipsilateral pelvic lymphocele at post-operative 6th month.

SECONDARY OUTCOMES:
Post-operative drainage | post-operative 3 days
  left and right post-operative drainage
lymphedema | post-operative 3 and 6 month
  lymphedema symptoms and sign at post-operative 3 and 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea